CLINICAL TRIAL: NCT00098501
Title: A Phase 1 Trial of CCI-779 in Combination With EKB-569, an EGFR Inhibitor, in Patients With Solid Tumors
Brief Title: CCI-779 and EKB-569 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01459; MC027C; NCI-6200; MAYO-MC027C; CDR0000398176; U01CA069912 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — EKB 569; temsirolimus; Sirolimus

ARMS (1):
- Arm I (Experimental): Patients receive oral EKB-569 on days 1-28 and oral CCI-779 on days 1-7 and 15-21.
  Interventions: Drug: pelitinib; Drug: temsirolimus

INTERVENTIONS:
Drug: pelitinib
  Other Names: EKB-569
Drug: temsirolimus — Given PO
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
This phase I trial is studying the side effects, best way to give, and best dose of CCI-779 and EKB-569 in treating patients with advanced solid tumors. Drugs used in chemotherapy, such as CCI-779, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. EKB-569 may stop the growth of tumor cells by blocking some of the enzymes needed for their growth. Giving CCI-779 together with EKB-569 may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of the combination of CCI-779 and EKB-569 in patients with advanced solid tumors.

II. Determine the toxicity of this regimen in these patients. III. Determine the response rate in patients treated with this regimen.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 3 treatment groups.

Group I: Patients receive oral EKB-569 on days 1-28 and oral CCI-779 on days 1-7 and 15-21.

Cohorts of 3-6 patients receive escalating doses of EKB-569 and CCI-779 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Group II: Patients receive oral EKB-569 at the MTD on days 4-28 of course 1 and days 1-28 of all subsequent courses and CCI-779 at the MTD on days 1-3 and 15-17.

Group III: Patients receive EKB-569 at the MTD as in group I and oral CCI-779 at the MTD on days 7-9 and 19-21 of course 1 and days 1-3 and 15-17 of all subsequent courses.

In all groups, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 30-42 patients (18-30 for group I, 6 for group II, and 6 for group III) will be accrued for this study within 1.35-1.75 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable solid tumor for which there is no known standard therapy that is potentially curative or capable of extending life expectancy
* No CNS metastases
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin normal
* AST ≤ 3 times upper limit of normal (ULN) (5 times ULN if liver involvement)
* Creatinine ≤ 1.5 times ULN
* No New York Heart Association class III or IV heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* Fasting cholesterol < 350 mg/dL
* Fasting triglycerides < 400 mg/dL
* No uncontrolled infection
* No seizure disorder
* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior biologic therapy
* No concurrent immunotherapy
* No concurrent prophylactic colony-stimulating factor therapy
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No other concurrent chemotherapy
* No concurrent oral contraceptives
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to > 30% of bone marrow
* No concurrent radiotherapy
* More than 7 days since prior CYP3A4 inducers
* No prior mTOR-targeting agents
* No prior epidermal growth factor receptor-targeting agents
* No concurrent antiretroviral therapy that induces or inhibits CYP3A4 for HIV-positive patients
* No other concurrent investigational agents
* No concurrent warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-10; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients | Up to 28 days
Number and severity of all adverse events per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 30 days after last dose of study treatment
  Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.

SECONDARY OUTCOMES:
Best response according to the Response Evaluation Criteria in Solid Tumors (RECIST) | Time from the start of the treatment until disease progression/recurrence, assessed up to 3 years
Time until any treatment related toxicity | Up to 3 years
Time until treatment related grade 3+ toxicity | Up to 3 years
Time until hematologic nadirs (white blood cells [WBC], absolute neutrophil count [ANC], platelets) | Up to 3 years
Time to progression | Up to 3 years
Time to treatment failure | Time from registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States